CLINICAL TRIAL: NCT01279408
Title: Prospective Observational Study Of Patients With Asymptomatic Centrally Located Advanced NSCLC Who Are Not Suitable For Curative Treatment
Brief Title: Observing Patients With Palliative Asymptomatic Centrally Located Advanced Non-small Cell Lung Carcinoma (NSCLC)
Status: Active, not recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: UHN REB 10-0484-CE
Record Dates: First submitted 2011-01-17; First posted 2011-01-19 (Estimated); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Non-small Cell Lung Carcinoma
Keywords: Palliative treatment; advanced non-small cell lung cancer; Patients with Asymptomatic Centrally Located Advance NSCLC who are palliative
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: None: Questionnaire Study — Patients enrolled in this study will have standard treatment as per the discretion of their attending physician. The only additional requirement is that they would be asked is to complete questionnaires

SUMMARY:
The aim of the study is to assess current practice within PROP & lung teams, for treating asymptomatic patients with centrally located non-small cell lung cancer (NSCLC), and to observe outcomes for those patients receiving immediate or deferred RT. This is a prospective cohort trial. Patients will be managed by immediate radiotherapy (RT) or a deferred approach according to physicians' individual current clinical practice. Baseline and follow-up data collection will be structured to focus on patient-reported measures to describe clinical outcomes in the two management groups. Indications for prescribing RT and dose fractionation schedules will also be collected. A new intervention will not be introduced during this trial. Instead, a follow-up regimen will be offered to both groups of patients, so that RT can be offered to the deferred group of patients if/when symptoms develop, and we can monitor symptoms/toxicities and QoL in both groups of patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC
* Central disease, as defined by tumour (either primary or nodal disease) arising or extending within a 2cm circumferential expansion from the centre of the trachea or within the zone of the proximal bronchial tree
* Disease is visible on thoracic CT (diagnostic or simulation)
* Asymptomatic from intra-thoracic tumour (may have background chest symptoms related to underlying COAD etc, but these symptoms must not have worsened due to tumour)
* Patient (due to age or co-morbidities) or tumour (due to locally advanced or metastatic disease) is not suitable for radical treatment (defined as surgery or RT dose >50Gy in 20 fractions or equivalent).
* Previous chemotherapy, thoracic RT or surgery is allowed
* RT to other metastases (e.g. brain, bone etc) is allowed

  •≥ 18 years of age
* Able to provide written informed consent

Exclusion Criteria:

* Intra-thoracic disease is peripheral only, not extending within 2cm of trachea/proximal bronchial tree
* Symptomatic from intra-thoracic NSCLC
* Histological diagnosis of small cell lung cancer, or malignant mediastinal lymphadenopathy from another malignancy (not NSCLC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Centrally Located Advanced NSCLC who are Asymptomatic and who are not Suitable for Curative Treatment
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
To determine the pattern of practice for management (immediate radiotherapy, deferred radiotherapy) of patients with ACLA-NSCLC, including reasons, timing and dose fractionation of lung/mediastinal RT | 6 years

SECONDARY OUTCOMES:
To describe the patient reported outcomes (symptoms, toxicities and quality of life measures) in patients with ACLA-NSCLC at 4 and 12 months | 6 years
To explore the relationship between utility and initial treatment decision (immediate versus deferred) | 6 years
To describe the disease status (as per CT imaging) at 4 months | 6 years
To describe the overall survival in patients with ACLA-NSCLC | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Wong, MBChB, Principal Investigator — University Health Network, Princess Margaret Hospital
Locations (1):
- University Health Network, Princess Margaret Hospital, Toronto, Ontario, Canada